CLINICAL TRIAL: NCT04111835
Title: HPV Testing In Polish POpulation-based Cervical Cancer Screening Program - a Randomized Healthcare Policy Trial
Brief Title: HPV Testing In Polish POpulation-based Cervical Cancer Screening Program.
Acronym: HIPPOPROJECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 28/2019; 28/2019/1/2020 (Other: Bioethics Committee of the Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland,)
Record Dates: First submitted 2019-09-19; First posted 2019-10-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; cervical screening; HPV testing
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exfoliative cytology/LBC (No Intervention): According to current Polish guidelines:
  ASC-US: repeat Pap testing in 6 months - current standard protocol
  LSIL - repeat Pap testing in 6 months or refer for colposcopy (by the decision of cytologist) - current standard protocol
  ASC-H and higher and all glandular lesions - refer for colposcopy - current standard protocol
  Colposcopy-targeted biopsies will be taken in agreement with national guidelines.
  If screening cytology is negative -> rescreening after 3 years.
- hrHPV molecular testing (Experimental): hrHPV-positive - reflex LBC:
  Abnormal reflex LBC (ASC-US or worse) -> colposcopy
  Normal reflex LBC -> repeat LBC in 6 months
  Positive - colposcopy
  Negative -> The CINtec PLUS Cytology and The QIASURE methylation test
  The CINtec PLUS Cytology Positive -> colposcopy Negative -> rescreen in 3 years
  The QIASURE methylation test Positive -> colposcopy Negative -> rescreen in 3 years
  Colposcopy-targeted biopsies will be taken in agreement with national guidelines.
  HPV-negative - rescreen in 5 years
  Interventions: Diagnostic Test: Offering an alternative cervical cancer screening method - hrHPV molecular testing.

INTERVENTIONS:
Diagnostic Test: Offering an alternative cervical cancer screening method - hrHPV molecular testing. — Women randomized to this screening strategy group will take a hrHPV molecular test.
  hrHPV-positive - reflex LBC:
  Abnormal reflex LBC (ASC-US or worse) -> colposcopy
  Normal reflex LBC -> repeat LBC in 6 months
  Positive - colposcopy
  Negative - rescreen in 3 years
  HPV-negative - rescreen in 5 years
  Arms: hrHPV molecular testing

SUMMARY:
The HIPPO PROJECT is a randomized healthcare study nested in the OCCSP in Poland. This project will assess the performance of the new screening test (HR HPV test) before its implementation in Poland.

DETAILED DESCRIPTION:
The study assumes randomized assumption of 33,000 women aged 30-59 to cytology or HR HPV test in a 1:1 ratio with age stratification (three strata: 30-39, 40-49 and 50-59 years).

Patients are recruited by the Cervical Cancer Prevention Clinic at the Department of Cancer Prevention at the Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw (main centre) and 8 more sites from distant regions of Poland (Lublin, Masovian, Silesian, Swietokrzyskie and West Pomeranian Voivodeship). All sites are selected through a tendering process and have to fulfil several criteria for inclusion into the project (active participation in the OCCSP, being certified for HPV testing with the chosen clinically validated hrHPV DNA assays)to obtain results representative for the entire country.

Gynaecological clinics:

Lublin Voivodeship:

* Non-Public Health Care Department MED -SPEC in Zamosc
* Plus Clinic in Zamosc
* Medical Center - Diagnostic in Lukow

Masovian Voivodeship:

* Medical Center - Diagnostic Siedlce, Kleeberg Street 2 Minsk Mazowiecki, Dąbrówki Street 2 Lukow, Krynka Street 1C Nur, Drohiczyńska Street 8, Sterdyn, Lipowa Street 1A, 08-320 Sterdyn Zelechow, Piłsudskiego Street 34 Strachowka, Norwida Street 6A Wierzbno, Wierzbno Street 88 Latowicz, Nowowiejska Street 34, Wielgolas
* Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw
* St. John Paul II Mazovian Provincial Hospital in Siedlce

Silesian Voivodeship:

* Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw on Gliwice
* SUPRA-MED in Bielsko-Biała
* SUPRA-MED in Wilkowice
* Gynecology and Obstetrics Clinic "K na Żeromskiego" in Wodzisław Slaski
* Medical Center in Rybnik
* Non-public Health Care JARO in Wodzisław Slaski
* Non-public Health Care EVA in Lubliniec
* SIKORNIK Clinic in Gliwice

Swietokrzyskie Voivodeship:

- Holy Cross Cancer Centre in Kielce

West Pomeranian Voivodeship:

* Non-public Health Care MULTIMED Gynecology and Obstetrics in Koszalin Koszalin, Monte Casino Street 13 Koszalin, Sw. Wojciecha Street 1 Koszalin, Kolejowa Street 71 Koszalin, Lelewela Street7 Bedzino Street 18
* "Hospital in Szczecinek"

Cytological&molecular laboratories

* Maria Sklodowska-Curie National Research Institute of Oncology; Roentgen Street 5, Warsaw, Armii Krajowej Street 15, 44-102 Gliwice (branch in Gliwice),
* Holy Cross Cancer Centre; Prezydent Stefan Artwinski Street 3, 25-734 Kielce,
* Medical Center - Diagnostic; Niklowa Street 9, 08-110 Siedlce,
* ALAB Laboratories; Stępinska Street 22/30, 00-739 Warsaw,
* Non-public Health Care Center MEDITEST Medical Diagnostics; Bronislawy Street 14D, 70-533 Szczecin,
* Non-public Health Care MULTIMED Gynecology and Obstetrics; Monte Casino Street 13, 75-414 Koszalin,
* Non-Public Health Care Department of Pathomorphology ALFAMED. Edward Cwierz, Maciej Cwierz; Jana Kilinskiego Street 78, 22a-400 Zamosc,
* Femina. Medical Centre; Klodnicka Street 23, 40-703 Katowice.

Colposcopy clinics

* Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw
* Non-public Health Care Center MEDITEST Medical Diagnostics in Szczecin
* Maria Sklodowska-Curie National Research Institute of Oncology in Gliwice
* Non-public Health Care MULTIMED Gynecology and Obstetrics
* St. John Paul II Mazovian Provincial Hospital in Siedlce
* Femina. Medical Centre in Katowice
* Holy Cross Cancer Centre in Kielce
* Medical Center - Diagnostic in Siedlce
* Non-Public Health Care Department of Pathomorphology ALFAMED. Edward Cwierz, Maciej Cwierz in Zamosc

The primary endpoint is the detection rate (DR) of histologically confirmed CIN2 or higher in each screening arm and detection rate ratio (DRR) of CIN2+ in HPV test vs cytology arm in intention-to-treat (ITT) analysis. Secondary endpoints include detection rate ratio of CIN1+, CIN3+ (including adenocarcinoma in situ) and invasive CC in both ITT and per-protocol (PP) analysis, restricted to women who adhered to the foreseen follow-up.

Other outcome measures are: (1) distribution of women by the screening test results; (2) referral rate for colposcopy; (3) compliance with referral for colposcopy; (4) positive predictive value of referral for colposcopy calculated for each screening test and separately by histology results (no CIN, CIN1, CIN2, CIN3, AIS, CIN2+, CIN3+, invasive cancer (squamous/adenocarcinoma)); (5) DR of histologically confirmed CIN2+ in patients with hrHPV positive test, two NILM LBCs six months apart and a positive CINtePlus Cytology and/or Qiasure test; (6) DRR of histologically confirmed CIN2+ after CINtec® PLUS Cytology test vs. QIASURE methylation test; (7) yield of use of CINtec® PLUS Cytology test vs. QIASURE methylation test in terms of detection rate of histologically confirmed CIN2+.

Additionally, biobanking of cytological samples taken from patients participating in the HIPPO Project is planned in Maria Sklodowska-Curie National Research Institute of Oncology for the purpose of potential future restrospective analyses if new cervical cancer screening technologies emerge.

The study was approved by the Bioethics Committee of National Research Institute of Oncology (ID: 28/2019/1/2020).

ELIGIBILITY:
Inclusion Criteria:

-women aged 30-59 with no screening Pap test within the preceding three years in the OCCSP and women with risk factors entitled to annual screening based on information from the SIMP and not tested within preceding 12 months (based on information from the screening database SIMP)

Exclusion Criteria:

-women with screening Pap test within the preceding three years in the OCCSP

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33000 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of histologically confirmed CIN2 or worse in each screening arm | 12 months after the date of the positive screening test
Detection rate ratio of CIN2+ in HPV test vs cytology arm (and detection rate ratios between the hrHPV test and cytology) | 12 months after the date of the positive screening test
  This is defined as:
  number of women with CIN2+ detected in the HPV arm/women screened by HPV
  ...........................................................................................................................
  number of women with CIN2+ detected in the cytology arm/women screened in with cytology

SECONDARY OUTCOMES:
Detection rate ratio of CIN1+, CIN3+ (including adeno-carcinoma-in-situ) and cervical cancer (ITT). | 12 months after the date of the positive screening test
Detection rate ratios of CIN2+ (and CIN1+, CIN3+, cancer) in the per-protocol analysis, restricted to women who adhered to the foreseen follow-up. | 12 months after the date of the positive screening test

OTHER OUTCOMES:
Distribution of women by the screening test results | 12 months after the date of the positive screening test
  This is for conventional cytology and LBC - according the modified Bethesda 2014 system used in the program. We will analyze the number of women due to the result of screening test in each arm.
Referral rate for colposcopy for each screening test | 12 months after the date of the positive screening test
  Analyses will be performed on data collected in SIMP. We will check the compliance on referral for colposcopy for each screening.
Positive predictive value of referral for colposcopy calculated for each screening test and separately | 12 months after the date of the positive screening test
  Histology: No CIN, CIN1, CIN2, CIN3, AIS, CIN2+, CIN3+, invasive cancer (squamous/adenocarcinoma).
Detection rates of histologically confirmed CIN2+ in patients with second negative LBC result | 12 months after the date of the positive screening test
  Detection rates of histologically confirmed CIN2+ in patients with second negative LBC result: after CINtec PLUS Cytology test and after QIASURE methylation test; detection rate ratio of histologically confirmed CIN2+ after CINTEC test vs after QIASURE methylation test
Yield of use of additional diagnostic tests in terms of detection rate of histologically confirmed CIN2+ | 12 months after the date of the positive screening test
  Number of women with histologically confirmed CIN2+ after CINtec test/number of women screened with HPV test
Yield of use of additional diagnostic tests in terms of detection rate of histologically | 12 months after the date of the positive screening test
  Number of women with histologically confirmed CIN2+ after QIASURE methylation test/number of women screened with HPV test

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Glinska P, Komerska K, Janik B, Olkowicz J, Jedrzejewska I, Macios A, Wieszczy P, Kaminski MF, Arbyn M, Nowakowski A. HPV testing in Polish population-based cervical cancer screening programme (HIPPO project)-study protocol of a randomised healthcare policy trial. BMC Cancer. 2023 Nov 17;23(1):1118. doi: 10.1186/s12885-023-11597-5. PMID 37978452